CLINICAL TRIAL: NCT02679495
Title: Positive Lifestyle Interventions for the Prevention of Gastric Pre-cancer and Cancer Occurrences in Patients With Chronic Atrophy Gastritis and Reccurence of Gastric Cancer After Endoscopic Resection
Brief Title: Lifestyle Intervention for Prevention of Gastric Neoplasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Lijun PENG, MD, Dr., Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015WS0366
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-05

CONDITIONS: Stomach Neoplasms
Keywords: early gastric cancer; lifestyle
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to lifestyle intervention group or the control group without lifestyle intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Active Comparator): A better lifestyle that are supposed to prevent gastric cancer occurrence are advised to patients. Measures includes dietary change and cessation of smoking and alcohol abuse. Behavioural and cognitive strategies from investigators are performed to patients to ensure adherence to established intervention.
  Interventions: Behavioral: Active measures of lifestyle modification
- No intervention (No Intervention): No meassures are taken to change life style of enrolled patients.

INTERVENTIONS:
Behavioral: Active measures of lifestyle modification
  Arms: Lifestyle intervention

SUMMARY:
The purpose of this study is to determine whether positive lifestyle interventions (diet modification and smoking cessation) are effective in the prevention of gastric pre-cancer and cancer occurrences and reccurence of gastric cancer after endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic atrophy gastritis proved by gastroscopy biopsy pathology or early gastric cancer patients who have recieved endoscopic resection
* have one or several bad lifestyle habits such as eating too much salt, eating too few fruits, smoking, drinking wine, and lack of sleep.

Exclusion Criteria:

* patients who refuse to change lifestyle according to the trial plan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
gastric caner occurrence | 4 years
  gastric cancer proved by gastroscopy biopsy

SECONDARY OUTCOMES:
All cause mortality | 5 years
gastric tissue DNA methylation change of selected genes | 4 years
  All patients have gastric biopsy through gastroscopy at the enrollment time and the last follow-up. DNA methylation status of selected genes are tested.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD, Study Chair — Shandong University
Locations (1):
- Linyi People's Hospital affiliated to Shandong University, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided